CLINICAL TRIAL: NCT06787105
Title: Fruquintinib in Patients With Metastatic Colorectal Cancer: A Prospective, Multicenter, Observational Study
Brief Title: Fruquintinib in Patients With Metastatic Colorectal Cancer
Acronym: FRUQUENT
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Takeda GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-100523
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: non-interventional; Fruzaqla; electronic QoL questionnaire; Real-world disease control rate; Later line; Fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
FRUQUENT is an observational study in Germany. The goal of the study is to evaluate how well Fruquintinib works to treat patients with metastatic colorectal cancer that have previously been treated with available standard therapies.

To this end, it will be analyzed how well patients respond to the therapy in the clinical routine. Further points of interest to the study are survival data, safety data, the use of medical care facilities, and the quality of life of patients treated with Fruquintinib.

Participants will be treated as decided by the treating physician and according to their routine practice.

DETAILED DESCRIPTION:
FRUQUENT is a prospective, multicenter, observational study in Germany, collecting real-world data of patients with metastatic colorectal cancer (mCRC) who receive fruquintinib according to the SmPC. The goal of the study is to analyze the effectiveness of the monotherapy with fruquintinib in adult patients with mCRC that have previously been treated with available standard therapies, including fluoropyrimidine, oxaliplatin-, and irintecan-based chemotherapies, anti-VEGF agents, and, if RAS wild-type, anti-EGFR agents. Moreover, the patients must have progressed on or be intolerant to treatment with either trifluridine/tipiracil or regorafenib.

All data for FRUQUENT will be obtained in routine clinical practice, allowing for a representative evaluation of the effectiveness of fruquintinib in a real-world setting. The study aims to recruit 150 patients in 50 practices (office based, oncology outpatient-centers or hospitals) to facilitate robust data.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Indication and decision for therapy with fruquintinib in accordance with the current German SmPC of fruquintinib as monotherapy for patients with mCRC.
* Prior treatment with available standard therapies, including fluoropyrimidine-, oxaliplatin-, and irinotecan based chemotherapies, anti VEGF therapy, and if RAS wild-type, anti EGFR therapy.
* Progression on or intolerance to treatment with either trifluridine/tipiracil and/or regorafenib.
* Other criteria according to current SmPC.
* Signed written informed consent.* * Patients are allowed to be enrolled up to 6 weeks after their first dose of fruquintinib. These patients cannot participate in the PRO assessments.

Exclusion Criteria:

* Participation in an interventional clinical trial (except follow-up) within 30 days prior to enrollment or start of treatment with fruquintinib, whatever comes first.
* Contraindications according to current SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with mCRC receiving fruquintinib in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Real-world disease control rate (RW DCR) | Start of treatment to end of treatment (avg. 6 months)
  The primary objective is to assess the effectiveness of fruquintinib in routine treatment. To this end, the real-world disease control rate will be analyzed, defined as the rate of complete response, partial response, or stable disease, either radiologically documented or clinically assessed by the treating physician.

SECONDARY OUTCOMES:
Best response | Start of treatment to end of treatment (avg. 6 months)
  Further effectiveness objective: Best response radiologically documented or clinically assessed by the treating physician.
Overall response rate (ORR) | Start of treatment to end of treatment (avg. 6 months)
  Further effectiveness objective: ORR is defined as proportion of patients with any response (partial or complete remission) overall, radiologically documented or clinically assessed by the treating physician.
Time to treatment failure (TTF) | Start of treatment to end of treatment (avg. 6 months)
  Further effectiveness objective: TTF is defined as the time from treatment start to discontinuation of treatment for any reason, including progression of disease, treatment toxicity, and death.
Time to next treatment (TTNT) | Start of treatment to start of subsequent antineoplastic therapy (max. 33 months)
  Further effectiveness objective: TTNT is defined as the interval from the start of fruquintinib treatment to initiation of the next line of therapy.
Progression-free survival (PFS) | Start of treatment to disease progression or death (max. 33 months)
  Further effectiveness objective: PFS is defined as the time from start of fruiquintinib treatment to disease progression or death from any cause.
Overall survival (OS) | Start of treatment to death (max. 33 months)
  Further effectiveness objective: OS is defined as the time from first administration of fruquintinib to death from any cause.
Adverse events (AEs) and serious adverse events (SAEs) according to NCI CTCAE | Start of treatment until 30 days after end of fruquintinib treatment (avg. 7 months)
  Safety objective: Incidence of (serious) AEs ((S)AEs) as characterized by type, frequency, severity and seriousness.
Adverse drug reaction (ADR) and serious adverse drug reactions (SADR) related to fruquintinib | Start of treatment to 30 days after end of fruquintinib treatment (avg. 7 months)
  Safety objective: Incidence of (serious) adverse drug reactions ((S)ADRs) as characterized by type, frequency, severity and seriousness.
Quality of life (QoL): Absolute values over time from baseline to end of study | Baseline to (individual) end of study (max. 33 months)
  Patient-Reported Outcome (PRO) objective: Evaluation of QoL by validated EORTC QLQ-C30 questionnaire during fruquintinib treatment and follow-up period using absolute values over time from baseline to end of study (EOS).
  The absolute values over time will be reported on the global health status / quality of life scale, functional scales (physical, role, emotional, cognitive, social) and symptom scales (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties). These scales are scored from 0 to 100. For the global health status/QoL, higher scores represent a higher QoL. For functional scales, higher scores indicate a higher/healthier level of functioning, while for symptom scales lower scores indicate a lower level of symptomatology/problems.
Quality of life (QoL): Change from baseline over time to end of study | Baseline to (individual) end of study (max. 33 months)
  Patient-Reported Outcome (PRO) objective: Evaluation of QoL by validated EORTC QLQ-C30 questionnaire during fruquintinib treatment and follow-up period using changes from baseline over time to end of study (EOS).
  The changes from the baseline over time will be reported on the global health status / quality of life scale, functional scales (physical, role, emotional, cognitive, social) and symptom scales (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties). These scales are scored from 0 to 100 and the change is reported as the difference between the scores at baseline and time of interest. For the global health status/QoL and functional scales, positive values indicate an improvement in quality of life while negative values indicate a deterioration in quality of life. For symptom scales, negative values indicate an improvement in symptom burden and positive values indicate an increase in symptom burden.
Quality of life (QoL): Time to definitive deterioration (TTD) | Baseline to (individual) end of study (max. 33 months)
  Patient-Reported Outcome (PRO) objective: Evaluation of QoL by validated EORTC QLQ-C30 questionnaire during fruquintinib treatment and follow-up period using the time to definitive deterioration (TTD).
  The time to definitive deterioration will be reported on the global health status / quality of life scale, functional scales (physical, role, emotional, cognitive, social) and symptom scales (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties). These scales are scored from 0 to 100 and the TTD is reported as the period of time until definitive deterioration for each scale.
Frequency of parameters affecting physicians' treatment decision making | Baseline
  Assessment of physicians' treatment decision making using the frequency of distinct parameters affecting therapy choice.
Fruiquintinib therapy duration | Start of treatment to end of treatment (avg. 6 months)
  Treatment reality objective: Duration of treatment with fruquintinib
Frequency of treatment modifications of fruquintinib therapy | Start of treatment to end of treatment (avg. 6 months)
  Treatment reality objective: Frequency of treatment modifications (treatment interruptions and dose reductions) with reasons
Frequency of prior therapies according to type, setting and substance | Baseline
  Treatment reality objective: Frequency of previous therapies (radiation, surgery, systemic with setting: adjuvant/ neoadjuvant/ palliative) and substances for prior systemic antineoplastic therapies.
Frequency of subsequent antineoplastic therapies | From date of end of fruquintinib treatment until end of study (max. 33 months)
  Treatment reality objective: Frequency of subsequent antineoplastic therapies including substances.
Duration of first subsequent therapy | From date of end of fruquintinib treatment until end of first subsequent therapy (max. 33 months)
  Treatment reality objective: Duration of first subsequent antineoplastic therapy after discontinuation of fruquintinib treatment.
Frequency of hospitalizations and emergency unit visits | Start of treatment to end of treatment (avg. 6 months)
  Medical resource utilization objective: Frequency of hospitalizations (planned and unplanned) and emergency unit visits during fruquintinib treatment.
Duration of hospitalizations | Start of treatment to end of treatment (avg. 6 months)
  Medical resource utilization objective: Duration of hospitalization during fruquintinib treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr. med. Sebastian Stintzing, Principal Investigator — Charité Campus Mitte Medizinische Klinik Hämatologie/Onkologie und Tumorimmunologie
Locations (1):
- Onkologische Schwerpunktpraxis, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No